CLINICAL TRIAL: NCT02385513
Title: A Randomised Controlled Trial Comparing Two-Dose Priming With the 10-Valent Pneumococcal Conjugate Vaccine at 6 and 10 Weeks to 6 and 14 Weeks in Nepali Children
Brief Title: PCV10 Immunogenicity Study Nepal 2015
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Patan Academy of Health Sciences (Other); University of Otago (Other); Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015/01
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Streptococcus Pneumoniae
Keywords: Immunogenicity
MeSH Terms: interventions — 10-valent pneumococcal conjugate vaccine; PHiD-CV vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6 + 10 weeks of age PCV10 priming (Active Comparator): 10 valent pneumococcal conjugate vaccine administered (PCV10) at 6 and 10 weeks of age with a booster at9 months of age and routine vaccines administered as per the Nepal EPI schedule
  Interventions: Biological: 10-valent pneumococcal conjugate vaccine
- 6 + 14 weeks of age PCV10 priming (Active Comparator): 10 valent pneumococcal conjugate vaccine administered (PCV10) at 6 and 14 weeks of age with a booster at 9 months of age and routine vaccines administered as per the Nepal EPI schedule
  Interventions: Biological: 10-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 10-valent pneumococcal conjugate vaccine
  Other Names: Synflorix

SUMMARY:
A single centre open-label, parallel group, randomised controlled trial, recruiting healthy Nepalese infants aged 40-60 days, who present to the immunisation clinic at Patan Hospital, Kathmandu, Nepal, randomised to receive a 10-valent pneumococcal conjugate vaccine (PCV10) at either;

1. 6+10 weeks and 9 months OR
2. 6+14 weeks and 9 months The study will enroll 152 healthy Nepalese infants in each treatment arm (304 in total). Demographic and clinical data will be collected on an electronic case report form to allow monitoring remotely. Participants will receive the study vaccine according to their allocated treatment arm in addition to their other routine vaccines. The investigators will collect 3 blood samples for analysis of serum antibody responses to the PCV10 vaccine serotypes throughout infancy (see Table 1). The data collected will be analysed in order to determine whether the 6+10 schedule is non-inferior to the 6+14 schedule in generating immune responses against the vaccine serotypes above the ≥0•35μg/mL threshold. These data will then be used to inform decision-making around augmenting the currently recommended 6+14 schedule to a 6+10 schedule in Nepal. The investigators will collect a nasopharyngeal swab at 2 time points to look at carriage of pneumococcus over time and to assess differences between the 2 groups. This is of critical importance because much of the programmatic impact of PCV is ultimately conferred by reductions in carriage at the community level and indirect effects resulting from that nasopharyngeal (NP) protection.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE Streptococcus pneumoniae is the predominant cause of bacterial pneumonia, meningitis and septicaemia in children worldwide, and disproportionately affects children from developing countries. Pneumococcal conjugate vaccines (PCVs) reduce pneumococcal disease burden by direct protection and by reducing nasopharyngeal carriage, thereby preventing transmission and inducing herd protection.

In Nepal, invasive pneumococcal disease (IPD) is responsible for a substantial disease burden in children. Surveillance conducted since 2005 at Patan Hospital, Kathmandu indicates the majority of IPD is due to serotypes 1, 5 and 14, and that the greater proportion occurs in late infancy and toddlerhood.7 Vaccine introduction began in January 2015 with PCV10. GAVI (Gavi, The Vaccine Alliance) has funded an impact assessment programme (including IPD, pneumonia, nasopharyngeal (NP) colonization and health economics), which is underway.

A randomised controlled trial conducted by investigators at Patan Hospital in collaboration with the Oxford Vaccine Group, using a 10-valent PCV, demonstrated a two-dose prime (at 6 and 14 weeks) and 9-month booster to have non-inferior immunogenicity at 18 weeks and 10 months and superior immunogenicity in early childhood (2-4 years of age) compared to a conventional three-dose priming only schedule (6, 10, and 14 weeks). This two-dose prime and boost schedule, with an 8 week interval between the priming doses, has been adopted as an acceptable schedule by the World Health Organization (WHO) and recommended in late 2014 by the Nepal Ministry of Health as a result of the study. However the WHO have also recommended the introduction of a single inactivated poliomyelitis virus vaccine at 14-weeks of age in order to mitigate the risk of outbreaks from vaccine derived serotype 2 poliomyelitis virus, to protect against serotype 2 poliomyelitis virus once countries switch to bivalent OPV (oral polio vaccine) from trivalent OPV, and to enhance immunogenicity to poliomyelitis vaccine serotypes 1 and 3. This has created a programmatic dilemma and concerns around vaccine coverage as a result of requiring three injections at the 14-week visit. Thus the Nepalese Ministry of Health, based on these concerns around public acceptance and feasibility have decided to move the second PCV10 priming dose from 14 weeks to 10 weeks of age. Given this decision it is essential to evaluate the immunogenicity of the intended schedule, comparing it to the schedule that has been shown to provide a level of immunogenicity that would predict substantial program impact on disease and colonisation. This importance is further increased given that the Nepal PCV10 impact study is currently underway and the limited data on two-dose priming schedules with a one-month interval between priming doses in other settings shows a reduction in immunogenicity.

Therefore this study will be undertaken in order to evaluate the immunogenicity of the 10-valent PCV priming at 6 and 10 weeks being implemented by the Nepal Ministry of Health, compared to priming at 6 and 14 weeks of age in healthy Nepali infants. In both groups a PCV10 booster will be given at 9 months of age.

Nepal Nepal is a low-income country in South Asia with a population of 25.8 million people and an estimated under 5 year mortality of 54/1000 live births. Access to health care varies considerably within the country, but as few as 18% of children under 5 years with pneumonia are taken to health care facilities. The capital city, Kathmandu, resides in a large valley, which in 2011 had a total population of about 1,744,240 people, with approximately 10% of these being children under 5 years of age.

The majority of children in Nepal receive immunisation through local government outpatient clinics. The national Expanded Programme of Immunisation (EPI )schedule being followed in Nepal currently includes Bacillus Calmette-Guérin (BCG) at birth, diphtheria-tetanus-whole cell pertussis-hepatitis B-Haemophilus influenzae type b (DTwP-HBV-Hib) and oral Polio (OPV) vaccines at 6, 10 and 14 weeks of age, IPV at 14 weeks of age, measles and rubella vaccine at 9 months of age, Japanese Encephalitis (JE) vaccine at 12-23 months of age (in endemic regions only; Kathmandu is one of these regions) and tetanus toxoid during pregnancy. Vaccine coverage is high in Nepal with over 90% of infants receiving DTP, by 14 weeks of age in the past 3 years. PCV10 vaccine at 6 and 10 weeks and a booster at 9 months of age was initiated in the new birth cohort only (i.e. no catch up program is being instituted ) as of January 2015 with roll-out beginning in the west of the country and expected to reach the whole of the country by late 2015.

The Patan Academy of Health Sciences and Patan Hospital will lead this study in Nepal. Patan Hospital is one of only two hospitals in Kathmandu with paediatric referral and inpatient services and is based in Lalitpur, in the south of the City. Over 300 children commence immunisation at the 'Under 14 clinic' in the Patan Hospital paediatric outpatient department each month.

Pneumococcal Disease in Kathmandu On-going surveillance of IPD serotypes has been occurring at Patan Hospital in Kathmandu since 2005, identifying all paediatric admission from whom pneumococcus is isolated from normally sterile body fluids. This programme was initially funded through PneumoADIP as part of the South Asia Pneumococcal Alliance (SAPNA) with extensive collection of clinical, radiological and laboratory data, demonstrating pneumococcus to be a significant cause of disease in children in Kathmandu, and is currently funded by the World Health Organisation.

Analysis of these data up until late 2012, show a predominance of non-vaccine serotypes in early infancy, followed by a shift towards vaccine serotypes, particularly serotype 1, in late infancy and into childhood. The finding of serotypes 1, 5 and, 14 to be the most frequent disease causing isolates is in keeping with data summarized in the Global Serotype Project which demonstrated serotype disease order of frequency in low-income countries was 14, 5, 1, 6B, 19F, 23F and 6A. The age distribution of vaccine type disease reinforces the importance of initiating vaccine coverage early in infancy such that early boosting at 9 months may be performed to maintain coverage into early childhood.

Immunogenicity of PCV10 in Kathmandu We previously conducted an open-label, parallel group, randomised controlled trial at Patan Hospital, Kathmandu, Nepal from June 2010 to November 2011 with follow-on between February and October 2013. In this study we compared the then WHO recommended PCV schedule of three priming doses in early infancy (6, 10, and 14 weeks) to a two-dose prime (6 and 14 weeks) and boost at 9 months of age. We demonstrated using the ten-valent PCV (PCV10) that the two-dose prime with booster at 9 months provided analogous immunogenicity to the three-dose prime schedule during early infancy, with improved protection through early childhood.

Global Polio Eradication Initiative Over the last decade the oral poliomyelitis vaccine (OPV) has been extremely efficacious in preventing wild-type polio disease across the world, including Nepal. The OPV used in the routine vaccine schedule contains three serotypes of weakened poliomyelitis virus (types 1, 2 and 3), and has facilitated the eradication of wild-type poliomyelitis in Nepal. On very rare occasions disease may occur as a result of circulating vaccine derived polio viruses (cVDPV), particularly of serotype 2. Thus, in countries such as Nepal, there is the situation where wild-type disease has been eradicated yet there remains a rare risk of vaccine derived disease outbreaks. This had led to the proposal to switch to a bivalent OPV (types 1 and 3), globally. This cannot happen however, unless populations are protected from type 2 disease through some other means. Furthermore the inactivated poliomyelitis vaccine (IPV), which is administered as an intramuscular injection, generates immunity using killed strains of the three poliomyelitis serotypes, and thus does not produce vaccine type disease or result in the emergence of cVDPV outbreaks. This has led the WHO to recommend the introduction of IPV in order to interrupt and mitigate the risk of cVDPV type 2 disease, prior to the phasing in of the bivalent OPV and cessation of OPV-type 2 use. In Nepal a single dose of the IPV at 14 weeks of age in addition to the routine schedule of trivalent OPV, has now been implemented (September 2014). Nepal was the first GAVI (Gavi The Vaccine Alliance) country to introduce IPV, and is ready to participate in the globally synchronized switch to bivalent OPV that will be coordinated by WHO in 2016 . IPV is given at 14 weeks of age; the proposed PCV10 schedule of 6 weeks, 14 weeks, and 9 months of age meant that children would receive three injections at 14 weeks of age (IPV, PCV10 and dose 3 of DTwP-HBV-Hib vaccine). The perception by the health care providers and the Ministry of Health is that this will not be acceptable and will lead to reduced vaccine coverage. Therefore the Nepal Ministry of Health has introduced in January 2015 PCV10 on a schedule of 6 weeks, 10 weeks, and 9 months of age.

Based on locally available IPD data and a prior immunogenicity study in Kathmandu, pneumococcal conjugate vaccination utilising PCV10 with two priming doses at 6 and 14 weeks followed by a 9-month booster has been demonstrated to be the WHO preferred schedule in comparison to a three-dose prime only schedule. However the WHO have also recommended the introduction of a single dose of IPV at 14 weeks of age in order to eradicate poliomyelitis serotype 2 vaccine strain disease. Local experts anticipate a poor uptake of vaccine at 14 weeks of age due to the increase in number of injections from one to three at this time-point. The Nepali government has thus suggested moving the 14 weeks PCV10 priming dose to the earlier 10 week time-point, however there are no immunogenicity data to support this decision. Therefore this study will aim to compare the immunogenicity of giving the two PCV10 priming doses at 6 and 10 weeks to that of 6 and 14 weeks. In addition this study will also evaluate the adverse event profile following the 14 weeks of age visit in the two treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 40-60 days at time of first study vaccination
* Parent/ guardian of participant is willing and able to give informed consent for participation in the study.
* In good general health as determined by:

  * medical history
  * physical examination
  * clinical judgment of the investigator
* Participants residing in Kathmandu
* Parents able (in the Investigators opinion) and willing to comply with all study requirements.

Exclusion Criteria:

* Parent/guardian unwilling or unable to give written informed consent to participate in the study
* Previous immunisation (excluding BCG, OPV, hepatitis B, measles or other government vaccine programme) or planned vaccination during the study period with vaccine not foreseen by this study protocol except influenza vaccine and oral polio vaccination as recommended locally.
* Premature birth (<37 weeks gestation)
* Previous hospital admission except where hospital stay would not compromise the study in the judgment of the investigator.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the vaccination, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 304 (Actual)
Dates: Start 2015-08-21 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
Non-inferiority (proportion of infants with serotype specific IgG ≥0•35μg/mL against pneumococcal vaccine serotypes) | 9 months
  The proportion of infants with serotype specific IgG ≥0•35μg/mL against pneumococcal vaccine serotypes at 9 months of age.

SECONDARY OUTCOMES:
Serotype proportions (proportion of infants who have PCV10 serotype-specific IgG ≥0•35μg/mL) | 9 months
  The proportion of infants who have PCV10 serotype-specific IgG ≥0•35μg/mL one month after the second priming dose of PCV10 and one month following the 9 month booster.
Serotype GMCs geometric mean concentrations (GMCs) of PCV10 serotype specific IgG) | 9 months
  The geometric mean concentrations of PCV10 serotype specific IgG one month following the second priming dose of PCV10, at 9 months of age, and one month following the 9 month booster for each of the two study groups.
Carriage (Serotype specific pneumococcal carriage) | 9 months
  Serotype specific pneumococcal carriage at age 6 weeks, 1 month following the second priming dose of PCV10 and at age 10 months.
Adverse events | 9 months
  The proportion of adverse events in each group in the week following the 14 weeks of age visit

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Kandasamy R, Gurung M, Thorson S, Yu LM, Galal U, Voysey M, Kelly S, Wahl B, Berbers G, Finnegan K, Ansari I, Paudel K, Murdoch DR, O'Brien KL, Kelly DF, Goldblatt D, Shrestha S, Pollard AJ. Comparison of two schedules of two-dose priming with the ten-valent pneumococcal conjugate vaccine in Nepalese children: an open-label, randomised non-inferiority controlled trial. Lancet Infect Dis. 2019 Feb;19(2):156-164. doi: 10.1016/S1473-3099(18)30568-1. Epub 2019 Jan 8. PMID 30635252